CLINICAL TRIAL: NCT01369862
Title: Randomised, Double-blind, Placebo-controlled, Phase I/II Study of Single Dose GHB16L2 Trivalent Influenza Vaccine in Healthy Adults
Brief Title: Study of Single Dose GHB16L2 Trivalent Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AVIR Green Hills Biotechnology AG (Industry)
Responsible Party: Thomas Muster PhD, CEO/CSO, AVIR Green Hills Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GHB-CS08
Record Dates: First submitted 2011-01-04; First posted 2011-06-09 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2011-08

CONDITIONS: Influenza, Human
Keywords: live attenuated flu vaccines; influenza A (H1N1); intranasal application; replication-deficient influenza virus
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPGNH buffer (Placebo Comparator): SPGNH buffer administration by liquid nasal spray
  Interventions: Biological: Placebo
- GHB16L2 (Experimental): Dose level ~7.0 log10 fTCID50/strain/person
  Interventions: Biological: GHB16L2

INTERVENTIONS:
Biological: GHB16L2 — A/Brisbane/59/07(H1N1)-like delNS1, A/Brisbane/10/07(H3N2)-like delNS1, B/Florida/04/06-like delNS1 virus reassortants
  Arms: GHB16L2
Biological: Placebo — SPGNH buffer
  Arms: SPGNH buffer

SUMMARY:
The purpose of this phase I/II trial is to evaluate safety and tolerability of a single dose of GHB16L2 administered by liquid nasal spray for vaccination against seasonal influenza virus infection. It is also performed to assess immunogenicity and pharmacokinetics (shedding).

DETAILED DESCRIPTION:
GHB16L2 intends to provide a novel vaccination for influenza virus infection. 80 healthy volunteers will be included at a ratio of 1:1 for GHB16L2 or placebo. GHB16L2 will be administered once on day 1. Follow-up visits will be performed on days 2, 8 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18-60 years
* Seronegative for one or two of the applied vaccine strains
* Low antibody titres for H1N1v
* Written informed consent to participate in this study
* For female volunteers of childbearing potential, provision of a history and current use of reliable contraceptive practices

Exclusion Criteria:

* Acute febrile illness (>37.3°C)
* Signs of acute or chronic upper or lower tract respiratory illnesses
* History of severe atopy
* Seasonal influenza vaccination in 2008/2009 and/or later seasons and/or pandemic influenza vaccination at any time
* Fever ≥38.0°C in the time period between the pre-screening visit and day 1
* Known increased tendency of nose bleeding
* Volunteers with clinically relevant abnormal paranasal anatomy
* Volunteers with clinically relevant abnormal laboratory values
* In female volunteers of childbearing potential, a positive urine pregnancy test
* Simultaneous treatment with immunosuppressive drugs incl. Corticosteroids (≥2 weeks) within 4 weeks prior to study medication application
* Clinically relevant history of renal, hepatic, GI, cardiovascular, haematological, skin, endocrine, neurological or immunological diseases
* History of leukaemia or cancer
* HIV or Hepatitis B or C seropositivity
* Volunteers who underwent rhino or sinus surgery, or surgery of another traumatic injury of the nose within 30 days prior to application of study medication
* Volunteers who have received antiviral drugs, treatment with immunoglobulins or blood transfusions, or an investigational drug within 4 weeks prior to study medication application
* Volunteers who have received anti-inflammatory drugs 2 days prior to study medication application
* Volunteers who are not likely to cope with the requirements of the study or with a significant physical or mental condition that may interfere with the completion of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From baseline to 30 days after end of study

SECONDARY OUTCOMES:
Seroconversion rates at day 29 | At day 29 (end of study)
  Seroconversion rates for HAI, MNA, IgA and IgG
Determination of the presence of GHB16L2 in mucosal samples (viral recovery/shedding) | 1 week post immunisation
Immune response factor at day 29 | At day 29 (end of study)
  Immune response factors for HAI, MNA, IgA and IgG

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Mossler C, Groiss F, Wolzt M, Wolschek M, Seipelt J, Muster T. Phase I/II trial of a replication-deficient trivalent influenza virus vaccine lacking NS1. Vaccine. 2013 Dec 16;31(52):6194-200. doi: 10.1016/j.vaccine.2013.10.061. Epub 2013 Oct 30. PMID 24183981